CLINICAL TRIAL: NCT02985138
Title: Comparison of Unilateral or Bilateral Fixation Using Pedicle Screws and TLIF in the Treatment of Lumbar Foraminal Stenosis
Brief Title: Comparison of Unilateral or Bilateral Fixation in the Treatment of LFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Xiaofei Cheng, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNPHO-161116
Record Dates: First submitted 2016-11-23; First posted 2016-12-07 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Lumbar Foraminal Stenosis
MeSH Terms: interventions — Pedicle Screws

ARMS (2):
- Unilateral fixation (Experimental): Patients undergoing TLIF and unilateral pedicle screw fixation
  Interventions: Procedure: TLIF and unilateral pedicle screw fixation; Device: Pedicle screw and cage
- Bilateral fixation (Active Comparator): Patients undergoing TLIF and bilateral pedicle screw fixation
  Interventions: Procedure: TLIF and bilateral pedicle screw fixation; Device: Pedicle screw and cage

INTERVENTIONS:
Procedure: TLIF and unilateral pedicle screw fixation — TLIF combined with posterior unilateral pedicle screw fixation
  Arms: Unilateral fixation
Procedure: TLIF and bilateral pedicle screw fixation — TLIF combined with posterior bilateral pedicle screw fixation
  Arms: Bilateral fixation
Device: Pedicle screw and cage — Pedicle screw and cage

SUMMARY:
TLIF is a popular lumbar fusion technique to perform interbody fusion. Pedicle screws providing initial stability have been developed to correct deformity, improve the rate of fusion and speed patient's postoperative recovery. Conventionally, bilateral pedicle screw fixation is a standard approach. Recently, studies have revealed that unilateral pedicle screw fixation provides equivalent clinical outcomes and fusion rates as compared with bilateral pedicle screw fixation in lumbar fusion. Meanwhile, the unilateral approach can reduce intraoperative blood loss and operating time. To our knowledge, few randomized controlled studies comparing unilateral versus bilateral instrumented TLIF in lumbar degenerative diseases have been reported. The purpose of this study is to compare clinical and radiographic outcomes in a series of patients with lumbar foraminal stenosis using instrumented TLIF with unilateral or bilateral pedicle screw fixation.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent.
* Patient is willing to be available for each examination scheduled over the study duration.
* Lumbar foraminal stenosis diagnosed by patient history, physical examination and image confirmation.
* Patient has symptoms referable to the stenosis level (low back pain, leg pain, tingling, numbness or weakness), which are relieved after a selective nerve root block.
* Has not responded to conservative treatment for a period of 3 months (e.g. bed rest, physical therapy, medication, manipulations, other).

Exclusion Criteria:

* Has systemic infection, highly communicable diseases, inflammatory or autoimmune disease (e.g. osteomyelitis, crohn's, rheumatoid arthritis, systemic lupus, gout, HIV/AIDS, active tuberculosis, venereal disease, active hepatitis).
* Has presence of active malignancy
* Has a history of severe allergy
* Has a significant medical history that, in the investigator's opinion, would not make them a good study candidate.
* Pregnant, or may become pregnant within follow-up period of study
* Has other spinal conditions that will interfere with clinical outcomes (e.g. spinal structural deformities, spinal fractures, ankylosing spondylitis, spinal tuberculosis, spinal infection, spinal tumors, symptomatic cervical spinal disease)
* Spondylolisthesis at the target level
* Has undergone previous lumbar surgery
* Has severe osteoporosis (T-score ≤ -3.5)
* BMI > 35kg/m2
* Has a diagnosis, which requires postoperative medication that interferes with fusion, such as steroids.
* Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, Ehlers-Danios syndrome or osteogenesis imperfecta)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) scores | 2 years postoperatively

SECONDARY OUTCOMES:
Adverse events related to procedure | 2 years postoperatively
Operative duration | 1 week postoperatively
Estimated blood loss | 1 week postoperatively
Length of hospital stay | 1 week after discharge
Spinal angles | 2 years postoperatively
  Radiographic parameters
Intervertebral space height | 2 years postoperatively
  Radiographic parameters
Foraminal height | 2 years postoperatively
  Radiographic parameters
Cost of treatment | 2 years postoperatively
Fusion rate | 2 years postoperatively
Oswestry Disability Index (ODI) | 2 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic Surgery, Shanghai Ninth People's Hospital, Shanghai, China